CLINICAL TRIAL: NCT05766189
Title: Utilizing Wastewater Surveillance Data in a Communications Campaign to Boost Vaccination Uptake in New York State: a Comparison-control Trial
Brief Title: Wastewater Surveillance to Boost COVID-19 Vaccine Uptake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BOOST-wastewater
Record Dates: First submitted 2023-02-15; First posted 2023-03-13 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Vaccination; Wastewater Surveillance

STUDY DESIGN:
Intervention Model Description: Difference-in-differences
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Receives communications on level of SARS-CoV-2 as identified in the wastewater
  Interventions: Behavioral: Wastewater vaccine prompts
- Comparison arm (No Intervention)

INTERVENTIONS:
Behavioral: Wastewater vaccine prompts — Social media communications showing levels of SARS-CoV-2 in wastewater
  Arms: Intervention arm

SUMMARY:
The goal of the study is to determine the effect of a communications campaign sharing wastewater surveillance data to influence vaccine uptake in a metropolitan and non-metropolitan environment. The study will be conducted in Onondaga and Cayuga counties in New York State. Individuals of all ages within the selected counties, located in metropolitan and non-metropolitan environments will receive the intervention. The evaluation study design is a comparison-control trial. The primary outcome measure is the proportion of vaccine-eligible individuals in the county that received the COVID-19 vaccine stratified by type of vaccine dosage and age group. Vaccination data will be aggregated to the county by the State Department of Health and shared with the research team. Wastewater data will be pulled from the wastewater surveillance network. A difference in differences analysis will be used to estimate the effect of the intervention on both the outcomes between intervention and comparison groups following the intervention, while adjusting for potential confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* None - county-level vaccine uptake - no direct interaction with people getting vaccines

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100000 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Vaccine uptake | up to 3 months
  Number of individuals receiving a booster COVID-19 vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Syracuse University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be gathered as part of the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT05766189/Prot_SAP_000.pdf